CLINICAL TRIAL: NCT02891668
Title: Hypothyroidism, Metabolism and Quality of Life - Focus on QOL, REE, Cognitive Function and Body Composition
Acronym: HYMAQ
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Bjarke Borregaard Medici, MD, PH.d. student, Herlev Hospital
Other Study IDs: Herlev-Hymaq
Record Dates: First submitted 2016-05-17; First posted 2016-09-07 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hypothyroidism
Keywords: Basal Metabolic rate; Quality of life; Resting energy expenditure; Insulin resistance; Cognitive Function; Body Composition
MeSH Terms: conditions — Hypothyroidism; Insulin Resistance | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hypothyroid: Levothyroxine treatment
  Interventions: Drug: Levothyroxine treatment
- Healthy volunteers: Matched on age and BMI 18 persons

INTERVENTIONS:
Drug: Levothyroxine treatment — Eltroxin/Euthyrox is part of the normal treatment for hypothyroidism, and the patient is treated equally, whether he/she participates or not.
  Other Names: Eltroxin, Euthyrox
  Groups: Hypothyroid

SUMMARY:
This project has the following primary aims:

The main objective is to delineate the association between changes in Resting energy expenditure (REE) and QOL in hypothyroid patients before and after one year of L-T4 treatment. To achieve this, the investigators plan to compare newly diagnosed hypothyroid patients soon after diagnosis before L-T4 therapy has been initiated after 6 months and after 1 year of treatment.

Primary endpoint is changes in REE compared to changes in QOL Secondary endpoint is changes in cognitive function and changes in body composition before and after one year of treatment and furthermore changes in insulin resistance following changes in body composition and free fatty acids (FFA).

DETAILED DESCRIPTION:
Subjects and Methods:

74 newly diagnosed hypothyroid patients of both genders and age between 20 and 75 years will be recruited from the out-patients clinic in Herlev and Gentofte Hospital and the general practitioners before start of substitution therapy. Participants will get an appointment immediately after diagnosis to avoid unnecessary delay of treatment. Shortly after diagnosis patients will undergo a test panel at the first experimental day, where patients arrives fasting.

* Psychological test using:

  * ThyPRO a thyroid-specific quality of life questionnaire(18),
  * Cognitive function by CALCAP® Abbreviated Test Battery,
  * Perceived cognitive deficit questionnaire (Perceived Deficits Questionaire)
  * Major Depression Inventory (MDI) questionnaire
* REE will be measured by a CCM-express calorimeter,
* DEXA-scan
* Blood samples will be taken and patients will be characterized through basic information.
* Insulin resistance will be assess through an oral glucose tolerance test (OGTT) At end of the first experimental day patients will start L-T4 therapy following national guidelines, with regular control of thyroid hormones to ensure optimal treatment. When patients are euthyroid and TSH is below 4 * 10-3 International Units pr liter (mU/l) patients will have blood samples monitored every 3 months for the rest of the trial.

After 6 and 12 months of treatment patients will undergo a similar experimental day and return to their general practitioner or outpatient clinic.

A control group of 18 matched healthy persons will undergo the first experimental day in the same way as the hypothyroid patients, except they do not start any kind of therapy and they only participate in the first experimental day.

ELIGIBILITY:
Inclusion Criteria:

* TSH > 10 mU/liter

Exclusion Criteria:

* Serious competing illness
* Pregnancy or planning to become pregnant
* Thyroidectomized patients
* Unable to speak and understand danish

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypothyroid patients.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life as measured with the ThyPro questionaire | 1 year
Changes in resting energy expenditure in KCal/day | 1 year

SECONDARY OUTCOMES:
Changes in Perceived Deficit Questionaire | 1 year
Changes in insulin resistance evaluated by MATSUDA index | 1 year
Changes in insulin resistance evaluated by HOMA index | 1 year
Changes in cognitive tests | 1 year
Changes in body composition asses through lean mass | 1 year
Changes in body composition asses through visceral adipose tissue | 1 year
Changes in body composition asses through fat mass | 1 year
Changes in free fatty acids | 1 year
Changes in cholesterol | 1 year
Changes in serum triglycerides | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bjarke Medici, MD, Principal Investigator — Bjarke Medici
Locations (1):
- Department of internal Medicine, Herlev Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Medici BB, Lerche la Cour J, Knop FK, Krakauer M, Michaelsson LF, Faber J, Watt T, Nygaard B. Predictors of Improvement in Quality of Life When Treating Hypothyroidism. J Thyroid Res. 2021 Jun 11;2021:5577217. doi: 10.1155/2021/5577217. eCollection 2021. PMID 34194721